CLINICAL TRIAL: NCT04685421
Title: Liposomal Bupivacaine Pharmacokinetic Study After Median Sternotomy Incision Infiltration in a Pediatric Cardiac Surgery
Acronym: CohortI-II
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI, Christopher Tirotta, no longer at NCH as of 5-26-23.
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Principal Investigator, Jenny Esteves, Research Regulatory Affairs, Nicklaus Children's Hospital f/k/a Miami Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020005RI
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Conditions
Keywords: pediatric cardiac surgery; median sternotomy incision

STUDY DESIGN:
Intervention Model Description: Study population of 30 pediatric cardiac surgery patients (ages 2 to 17_cohort I) undergoing elective operations between the ages of two through seventeen years. Cohort II (Ages 2 < 6)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Liposomal Bupivacaine PK (Experimental): Liposomal Bupivacaine PKs collections up to 96 hours on children from 2 to 17 years in pediatric cardiac surgeries.
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine liposome — Liposomal Bupivacaine PKs collections up to 96 hours on children from 2 to 17 years in pediatric cardiac surgeries.
  Other Names: Bupivacaine liposome PKs

SUMMARY:
The purpose of the study is to determine the plasma concentration of bupivacaine at various time points after Exparel (bupivacaine liposome injectable suspension, Pacira Pharmaceuticals, Inc., Parsippany, NJ) is injected subcutaneously for median sternotomy incisions in pediatric cardiac surgery patients.

DETAILED DESCRIPTION:
To determine the pharmacokinetic profile and peak bupivacaine plasma concentration with the use of an Exparel/bupivacaine mixture in children ages two through seventeen (Cohort I). Cohort II covers ages 2 <6. We will be collecting blood samples at different times during 96 hours or until the patient is discharged from the hospital. There will be two different groups participating in the study alternating the times in which the blood samples will be collected. We hypothesize that peak plasma concentration will be significantly less than the toxic plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* Every elective pediatric surgery patient ages two through seventeen years old, inclusive.

Exclusion Criteria:

* Patients who fall outside of the age range for the study will be excluded. -Patients known to have had an anaphylactic or severe reaction to the drug or its components will not be enrolled. Any with Significant Liver Disease will also be excluded. Emergency patients will be excluded. Pregnant patients will be excluded.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Bupivacaine-Exparel levels | 96 hours
  To determine plasma bupivacaine levels after the use of Exparel 1.3% admixed with 0.25% bupivacaine and 0.9% Normal Saline in pediatric cardiac surgery patients ages two through seventeen years of age (Cohort I). Cohort II covers ages 2 < 6.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Tirotta, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nickalus Children's Hospital f/k/a Miami Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified will be posted in website.
Supporting Information: Study Protocol, ICF
Time Frame: one year after study closure
Access Criteria: Information will be provided by request to the PI

REFERENCES:
- [Background] Chughtai M, Sultan AA, Hudson B, Goodwin RC, Seif J, Khlopas A, Bena J, Jin Y, Gurd DP, Kuivila TE, Ballock RT. Liposomal Bupivacaine Is Both Safe and Effective in Controlling Postoperative Pain After Spinal Surgery in Children: A Controlled Cohort Study. Clin Spine Surg. 2020 Dec;33(10):E533-E538. doi: 10.1097/BSD.0000000000000996. PMID 32324672
- [Background] Crowley JS, McLean P, Gabriel RA, Cronin B, Hsieh S, Englar K, Said E, Lance S, Gosman A. The Association of Liposomal Bupivacaine on Opioid Consumption in the Pediatric Alveolar Cleft Population. J Craniofac Surg. 2020 Jun;31(4):1078-1081. doi: 10.1097/SCS.0000000000006310. PMID 32195834
- [Background] Cohen B, Glosser L, Saab R, Walters M, Salih A, Zafeer-Khan M, Rivas E, Zhang K, Schacham NY, Chodavarapu P, Essber H, Chelnick D, Raza S, Hanline C, Khoshknabi D, Yang D, Seif J, Chhabada S, Turan A. Incidence of adverse events attributable to bupivacaine liposome injectable suspension or plain bupivacaine for postoperative pain in pediatric surgical patients: A retrospective matched cohort analysis. Paediatr Anaesth. 2019 Feb;29(2):169-174. doi: 10.1111/pan.13561. Epub 2018 Dec 31. PMID 30521078
- [Background] Cloyd C, Moffett BS, Bernhardt MB, Monico EM, Patel N, Hanson D. Efficacy of liposomal bupivacaine in pediatric patients undergoing spine surgery. Paediatr Anaesth. 2018 Nov;28(11):982-986. doi: 10.1111/pan.13482. Epub 2018 Sep 11. PMID 30207019
- See also: Nicklaus Children's Hospital — http://www.nicklauschildrens.org